CLINICAL TRIAL: NCT07012356
Title: Does The Type of Hr-HPV and Multiple HPV Carrier Status Increase The Effectiveness of The Colposcopy in Diagnosing Preinvasive Lesions Using The Swede Score and The 2011 IFCPC Nomenclature?
Brief Title: Does Hr-HPV Status Influence the 2011 IFCPC Nomenclature and Swede Score's Capacity to Diagnose Precancerous Lesions?
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Cemre Alan, Principal investigator, Necmettin Erbakan University
Other Study IDs: 2024/4991
Record Dates: First submitted 2025-04-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Colposcopy; HPV; HSIL
Keywords: colposcopy; HPV; HSIL

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hr-HPV positive women who undergo colposcopy: Women referred for colposcopy to the gynecologic oncology outpatient clinic of a university hospital between June 2024 and November 2024 for high-risk HPV carriers.

SUMMARY:
Purpose: This study aims to examine the effectiveness of the Swede score and 2011 IFCPC Nomenclature in hr-HPV carriers and evaluate diagnostic sensitivity and specificity according to hr-HPV types and multiple HPV carrier status.

Methods: This study included 95 women with high-risk HPV. Colposcopic findings were scored using the Swede Score and the 2011 IFCPC system to predict pathology. Accuracy, sensitivity, specificity, PPV and NPV were calculated.

DETAILED DESCRIPTION:
This prospective study aims to examine the effect of 2011 IFCPC terminology, Swede score, and HPV type on the prediction of cervical precancerous lesions or cervical cancer in patients referred for colposcopy to the gynecologic oncology outpatient clinic of a university hospital between June 2024 and November 2024 for high-risk HPV carriers. An expert colposcopist evaluated all referred patients.

Sample size: a sample size of 95 has been determined using the formula n = [(Zα)2 × p(1 - p)] / e2, with allowable error of 7%, and p value = 0.781, derived from the study done by Shojaei et al.

n = [(1.645)2 × 0.781(1-0.781)] / 0.072. z score was used for 90% CI. 95 women underwent colposcopic examination and biopsy of at least one quadrant. All patients were positive for at least 1 type of high-risk HPV. Colposcopic features were assessed using the Swede Score and the IFCPC system 2011. The same colposcopist carried out all colposcopies and scoring.

All data collected were statistically analyzed using SPSS statistical software (version 22, Chicago, IL, USA). The Kappa coefficient was calculated to assess inter-rater agreement, while Spearman's rho was used to analyze the relationship between positively paired samples. Concerning the Swede score, the investigators have assessed the effectiveness of using cut-off values of 5 and 7 to identify HSIL. The investigators also examined whether the sensitivity and specificity of these scoring systems changed when they were evaluated together with data on the HPV type and multiple hr-HPV carrier status of the patients.

Descriptive statistics were conducted to analyse the demographic characteristics of the participants. Accuracy, sensitivity, specificity, PPV, NPV, and 95% confidence intervals were calculated by the SPSS program. The AUC construction was calculated from the sensitivity and specificity of the 2011 IFCPC Nomenclature and Swede score. A p-value < 0.05 was used for all statistical tests to indicate a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Women who are positive for at least 1 type of high-risk HPV.
* Women with high-risk HPV and subjective symptoms such as post-coital bleeding or prolonged leucorrhoea were included in the study.

Exclusion Criteria:

* Women with normal colposcopy findings, as defined by both the 2011 IFCPC system and the Swede score
* Pregnant women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a study about effectiveness of colposcopy, so female participants who have cervix uteri can be involved in the study. Women without a cervix (due to a n operation or congenital) are excluded.
Study Population: patients referred for colposcopy to the gynecologic oncology outpatient clinic of a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
The comparison of diagnostic power of the Swede Score and 2011 IFCPC Nomenclature in patients with hr-HPV | 6 months
  Thestudy aims to compare of diagnostic accuracy of the Swede Score and 2011 IFCPC Nomenclature in patients with hr-HPV. Receiver operating curves (ROC) are used for this comparison.

SECONDARY OUTCOMES:
The effectiveness of the Swede score and IFCPC in hr-HPV carriers according to HPV types and multiple HPV carrier status | 6 months
  This study aims to evaluate if effectiveness of the Swede score and IFCPC Nomenclature is changed by patients' HPV types and multiple HPV carrier status. For the IFCPC Nomenclature, major findings and for the Swede score, values of 5 and above were evaluated in terms of diagnosing HSIL lesions.
The effectiveness of the Swede score in hr-HPV carriers | 6 months
  This prospective study aims to examine the effect of Swede score on the prediction of cervical precancerous lesions or cervical cancer in patients referred for colposcopy to the gynecologic oncology clinic of a hospital between June 2024 and November 2024 for high-risk HPV carriers. ROC were used to show the correlation of the scoring system with final pathology results.The values of 5 and above were evaluated in terms of diagnosing HSIL lesions.
  Swede Score 0 1 2 Aceto uptake Zero or transparent Milky Opaque white Margins/Surface Diffuse Sharp, geographical satellites Sharp, surface level Vessels Fine and regular Absent Coarse or atypical Lesion size <5mm 5-15mm or 2 quadrants >15mm or 3-4 quadrants Iodine staining Brown Yellow Distinct yellow
The effectiveness of the 2011IFCPC Nomenclature in hr-HPV carriers | 6 months
  This prospective study aims to examine the effect of 2011 IFCPC terminology on the prediction of cervical precancerous lesions or cervical cancer in patients referred for colposcopy to the gynecologic oncology outpatient clinic of a university hospital between June 2024 and November 2024 for high-risk HPV carriers. Receiver Operating Curves (ROC) were used tos how the correlation of the scoring system with final pathology results. For the IFCPC Nomenclature, major findings were evaluated in terms of diagnosing HSIL lesions.
  Major findings in 2011 IFCPC Nomenclature are defined as; dense acetowhite epithelium, rapid appearance of acetowhitening, cuffed crypt, and coarse mosaic with sharp or inner border.

CONTACTS AND LOCATIONS:
Overall Officials: Cemre Alan, Dr, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alan M, Gunyeli I, Gultekin M, Sanci M, Yuce K. Correlation of Swede score colposcopy scoring system and histopathological results in patients with high-risk HPV infection other than HPV16 and 18. Int J Gynecol Cancer. 2020 Jan;30(1):35-40. doi: 10.1136/ijgc-2019-000932. Epub 2019 Dec 1. PMID 31792083
- [Result] Rahman Z, Yadav G, Tripathi U. The Diagnostic Efficacy of Swede Score for Prediction of Pre-invasive Cervical Lesions: A Prospective Hospital-Based Study. J Obstet Gynaecol India. 2020 Dec;70(6):497-502. doi: 10.1007/s13224-020-01344-2. Epub 2020 Jul 4. PMID 33417628
- [Result] Li Y, Duan X, Sui L, Xu F, Xu S, Zhang H, Xu C. Closer to a Uniform Language in Colposcopy: Study on the Potential Application of 2011 International Federation for Cervical Pathology and Colposcopy Terminology in Clinical Practice. Biomed Res Int. 2017;2017:8984516. doi: 10.1155/2017/8984516. Epub 2017 May 25. PMID 28626767
- [Result] Fan A, Wang C, Zhang L, Yan Y, Han C, Xue F. Diagnostic value of the 2011 International Federation for Cervical Pathology and Colposcopy Terminology in predicting cervical lesions. Oncotarget. 2018 Jan 8;9(10):9166-9176. doi: 10.18632/oncotarget.24074. eCollection 2018 Feb 6. PMID 29507681
- [Result] Li J, Wang W, Yang P, Chen J, Dai Q, Hua P, Liu D. Analysis of the agreement between colposcopic impression and histopathological diagnosis of cervical biopsy in a single tertiary center of Chengdu. Arch Gynecol Obstet. 2021 Oct;304(4):1033-1041. doi: 10.1007/s00404-021-06012-y. Epub 2021 Mar 8. PMID 33683424
- [Result] Qin D, Bai A, Xue P, Seery S, Wang J, Mendez MJG, Li Q, Jiang Y, Qiao Y. Colposcopic accuracy in diagnosing squamous intraepithelial lesions: a systematic review and meta-analysis of the International Federation of Cervical Pathology and Colposcopy 2011 terminology. BMC Cancer. 2023 Feb 23;23(1):187. doi: 10.1186/s12885-023-10648-1. PMID 36823557
- [Result] Zhang B, Hong S, Zhang G, Rong F. Clinical application of the 2011 IFCPC colposcope terminology. BMC Womens Health. 2021 Jun 24;21(1):257. doi: 10.1186/s12905-021-01395-1. PMID 34167543
- [Result] Bowring J, Strander B, Young M, Evans H, Walker P. The Swede score: evaluation of a scoring system designed to improve the predictive value of colposcopy. J Low Genit Tract Dis. 2010 Oct;14(4):301-5. doi: 10.1097/LGT.0b013e3181d77756. PMID 20885156
- [Result] Quaas J, Reich O, Frey Tirri B, Kuppers V. Explanation and Use of the Colposcopy Terminology of the IFCPC (International Federation for Cervical Pathology and Colposcopy) Rio 2011. Geburtshilfe Frauenheilkd. 2013 Sep;73(9):904-907. doi: 10.1055/s-0033-1350824. PMID 24771940
- [Result] Bornstein J, Bentley J, Bosze P, Girardi F, Haefner H, Menton M, Perrotta M, Prendiville W, Russell P, Sideri M, Strander B, Tatti S, Torne A, Walker P. 2011 colposcopic terminology of the International Federation for Cervical Pathology and Colposcopy. Obstet Gynecol. 2012 Jul;120(1):166-72. doi: 10.1097/AOG.0b013e318254f90c. PMID 22914406
- [Result] Wang P, Gao D, Yu X, Zhu G. Value of high-risk human papillomavirus detection combined with colposcopy in the diagnosis of cervical cancer and precancerous lesions. Oncol Lett. 2024 Feb 29;27(4):185. doi: 10.3892/ol.2024.14318. eCollection 2024 Apr. PMID 38476208
- [Result] Campos PL, Guimaraes ICCDV, Fialho SCAV, Martins CAO, Rodrigues FR, Velarde LGC, Monteiro DDSA. Association of Swede Score and 2011 IFCPC Nomenclature in Women with Abnormal Cytology. Rev Bras Ginecol Obstet. 2022 Oct;44(10):938-944. doi: 10.1055/s-0042-1751074. Epub 2022 Nov 29. PMID 36446560
- [Result] Li M, Du X, Lu M, Zhang W, Sun Z, Li L, Ye M, Fan W, Jiang S, Liu A, Wang M, Meng Y, Li Y. Prevalence characteristics of single and multiple HPV infections in women with cervical cancer and precancerous lesions in Beijing, China. J Med Virol. 2019 Mar;91(3):473-481. doi: 10.1002/jmv.25331. Epub 2018 Nov 13. PMID 30281807